CLINICAL TRIAL: NCT04542252
Title: An Open-label, Randomized, Crossover Study to Evaluate the Drug Interaction of Coadministered Cyclosporine on the Pharmacokinetics and Safety of Intravenous Administration of SyB V-1901 in Japanese Healthy Subjects
Brief Title: Drug-Drug Interaction Study of Intravenous Administration of SyB V-1901 and Cyclosporine in Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BCV-HV01
Record Dates: First submitted 2020-08-29; First posted 2020-09-09 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): SyB V-1901 alone, Simultaneous administration of SyB V-1901 and cyclosporine, Coadministration of cyclosporine at 2 hours after the completion of SyB V-1901 infusion
  Interventions: Drug: SyB V-1901; Drug: Cyclosporine
- Group 2 (Experimental): Simultaneous administration of SyB V-1901 and cyclosporine, SyB V-1901 alone, Coadministration of cyclosporine at 2 hours after the completion of SyB V-1901 infusion
  Interventions: Drug: SyB V-1901; Drug: Cyclosporine

INTERVENTIONS:
Drug: SyB V-1901 — SyB V-1901 10 mg via IV infusion for 2 hours
Drug: Cyclosporine — 200 mg Capsule

SUMMARY:
To evaluate the effect of coadministered cyclosporine on the pharmacokinetics of brincidofovir following simultaneous administration of SyB V-1901 with cyclosporine, or coadministration of cyclosporine at 2 hours after the completion of SyB V-1901 infusion in healthy adult subjects

DETAILED DESCRIPTION:
This study is an open-label, randomized and crossover study designed to evaluate the effect of cyclosporine on the pharmacokinetics of SyB V-1901. Healthy adult subjects will receive an IV dose of SyB V-1901 alone, simultaneous administration of SyB V-1901 with cyclosporine, and coadministration of cyclosporine at 2 hours after completion of SyB V-1901 infusion. Eligible subjects will be randomized to one of two groups, to receive the treatment sequence of assigned group.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy adult male aged between 20 to 55 years at informed consent
* BMI from 18 to 32 kg/m2 with a body weight of ≥ 50 kg
* Creatinine Clearance ≥ 60 mL/min at screening
* Judged to be in good general health, based on the review of medical history and the screening and Pre-Day1 examination

Main Exclusion Criteria:

* Positive for HIV antibody, or HBs antigen, or HCV antibody at the screening or within 6 months prior to the start of screening
* Have a history of infection of SARS-CoV-2, or subjects who have close contact with infected patients of SARS-CoV-2 within 2 weeks prior to screening or visit to epidemic area of SARS-CoV-2 infection in outside of Japan or have close contact with person who visit to epidemic area of SARS-CoV-2 infection within 2 weeks prior to screening
* Positive for SARS-CoV-2 polymerase chain reaction (PCR) in lower respiratory tract specimens, nasopharyngeal swabs or saliva and so on at screening or have a fever ≥ 37.5 °C and respiratory symptoms
* Have a history of drug abuse or alcohol dependence within 2 years prior to the start of screening
* Have a history of gastrointestinal disorders or cholecystectomy etc., which could interfere with the absorption of cyclosporine or could interfere with normal gastrointestinal anatomy or motility, but except for uncomplicated appendectomy.
* Have a history or symptoms of cardiovascular disease, including but not limited to coronary artery disease, hypertension, congestive heart disease, and clinically significant cardiac disorder.
* Have a history of hematological disorders or have a risk of gastrointestinal bleeding
* Have a history of chronic liver disease or hepatic impairment, including but not limited to alcoholic liver disease, chronic viral hepatitis, autoimmune hepatitis, steatosis or hemochromatosis.
* Have increased Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) greater than ULN at screening or Pre-Day1
* History of Gilbert's syndrome or increased total bilirubin greater than 1.5x the upper limit of the normal range at screening or Pre-Day1
* Have symptoms of infection within 2 weeks prior to Pre-Day1
* Have clinically significant abnormal hemoglobin at the screening or Pre-Day1, or a clinically significant iron deficiency
* Have a history of blood donation or had clinically significant blood loss within 30 days prior to Day 1, or platelet/plasma donation within 7 days prior to Day 1
* Have received any investigational drug, or device within 30 days prior to Day1
* History of tobacco- or nicotine-containing product use within 6 months prior to Day1

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of brincidofovir (BCV) | From initiation of SyB V-1901 administration though 16 days
Area under the plasma concentration versus time curve (AUC) of BCV | From initiation of SyB V-1901 administration though 16 days

SECONDARY OUTCOMES:
Cmax of cidofovir (CDV) | From initiation of SyB V-1901 administration though 16 days
AUC of CDV | From initiation of SyB V-1901 administration though 16 days
Cmax of Intercellular Cidofovir diphosphate (CDV-PP) in Peripheral Blood Mononuclear Cells (PBMCs) | From initiation of SyB V-1901 administration though 18 days
AUC of Intercellular CDV-PP in PBMCs | From initiation of SyB V-1901 administration though 18 days
Cmax of cyclosporine in blood | From initiation of cyclosporine administration though 16 days
AUC of cyclosporine in blood | From initiation of cyclosporine administration though 16 days
Number of subjects with adverse events (AE) | Follow up 22 days post dose
Number of subjects with severity of AEs | Follow up 22 days post dose
Number of subjects with abnormal findings for laboratory parameters | Follow up 22 days post dose
Number of subjects with abnormal findings for blood pressure | Follow up 22 days post dose
Number of subjects with abnormal findings for respiratory rate | Follow up 22 days post dose
Number of subjects with abnormal findings for heart rate | Follow up 22 days post dose
Number of subjects with abnormal findings for temperature | Follow up 22 days post dose

OTHER OUTCOMES:
Genotype of CYP4F2 | Pre-Day1
Genotype of OATP1B1 | Pre-Day1

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Yoshida, Study Director — SymBio Pharmaceuticals
Locations (1):
- Research Site, Hachioji-shi, Tokyo, Japan